CLINICAL TRIAL: NCT04859413
Title: Frequency Analysis of the Ultrasound Images in Rotator Cuff Tendon
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202102043RINA
Record Dates: First submitted 2021-04-19; First posted 2021-04-26 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Rotator Cuff Injuries
Keywords: ultrasonography; rotator cuff tendon
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- the young group: healthy participants age between 20 and 40
- the elder group: healthy participants age over 60

SUMMARY:
Previous studies used spatial frequency analysis of tendon ultrasound images and considered that the parameters can reflect the micro-structure of the tendon. In this study, we try to recruit and analysis the rotator cuff tendon in healthy adults with different ages and different equipment to explore the the normal range and differences of spatial frequency parameters. The hypotheses of this study are (1) the young and the elderly would have significantly different spatial frequency value; and (2) there would be significant different results between different equipment.

DETAILED DESCRIPTION:
Tendons are hierarchical fibrous tissues. The speckle signals of ultrasonic images have parallel stripes arranged along the long axis of the tendon, reflecting the arrangement of collagen fiber bundles in the tendon. The micro-structure of tendons can be quantified by analyzing the speckle pattern of ultrasonic images. A research team used fast Fourier transform to convert ultrasound images of tendons into two-dimensional spatial frequency spectra, and used linear discriminate analysis to calculate multiple spatial frequency parameters. The results indicated that there were 5 parameters with the highest accuracy in discriminating Achilles tendinopathy. There is a significant difference in the spectrum frequency parameters of whether the tendon was loaded and whether there was a tendinopathy tendon. Past studies using spatial frequency analysis in patients with shoulder pain, and they found that there was no significant difference between the asymptomatic control group and shoulder pain patients. The risk factors of rotator cuff tendon injury is related advanced age, dominant hand, and repeated overhead activities. Therefore, in this study, we will recruit participants of different ages and investigate the results of spatial frequency analysis of bilateral shoulders ultrasound images. The aim of this study is to know whether these factors may affect the micro-structure of the rotator cuff tendons and establish the reference norm of spatial frequency analysis parameters in those without obvious tendon degeneration or injury. In addition, we aim to compare the differences between spectrum analysis parameters with several instruments by using different ultrasonic equipment. This study could provide a reference for the clinical application of spatial frequency analysis in tendon ultrasound images.

ELIGIBILITY:
Inclusion Criteria:

* (1) age between 20-40 or age over 60;
* (2) no bilateral shoulder pain or discomfort within six months;
* (3) no past diagnosis in shoulder or upper extremities.

Exclusion Criteria:

* (1) fracture of upper extremities before;
* (2) be diagnosed as neck radiculopathy, central nervous system lesion of brain, or peripheral nervous system lesion of upper extremities;
* (3) rheumatoid arthritis or autoimmune disease;
* (4) have received any shoulder injection or surgery;
* (5) tendon tear in shoulder sonograms.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: adults from NTUH rehabilitation outpatient department, from NTU, or adults in connection with colleagues in the NTUH rehabilitation department or School and Graduate Institute of Physical Therapy in Collage of Medicine of NTU.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-04 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
spatial frequency analysis parameters | Day 1
  spatial frequency analysis in the ultrasound images of rotator cuff tendon

CONTACTS AND LOCATIONS:
Overall Officials: Chao Yuan-Hung, PhD, Principal Investigator — National Taiwan University Hospital